CLINICAL TRIAL: NCT03923491
Title: A Home-based Video and Motivational Interviewing Intervention to Improve Preschoolers Diet Quality and Parental Food Parenting Practices
Brief Title: A Home-based Intervention to Improve the Diet Quality of Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Brown University (Other); University of Connecticut (Other)
Responsible Party: Principal Investigator, Alison Tovar, Associate Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R34HL140229-01A1 (NIH)
Record Dates: First submitted 2018-08-14; First posted 2019-04-22 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Diet Modification
MeSH Terms: interventions — Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Intervention vs. Attention Control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Feeding, Healthy Eating (Experimental): The experimental arm will receive three home over the first three months of the intervention.Visits will be conducted by a community health worker (CHW) trained in Motivational Interviewing. The home visits will include video-feedback on a meal; in-home cooking demonstrations; tailored text-messages, and mailed materials. During the last three months of the intervention, CHW will conduct monthly phone calls, together with mailed materials and text messages. The intervention will be tailored for families based on the child's appetitive traits and eating behaviors.
  Interventions: Behavioral: Healthy Feeding, Healthy Eating
- Reading and Readiness (Active Comparator): The Reading and Readiness group will receive information on school readiness promotion. Materials will be adapted and delivered by the community health worker (CHW) with a similar dose and schedule as the intervention group (three home visits and three phone calls). During the home visits, the CHW will show a video that models early childhood caregiver-child activities and demonstrates simple methods to interact with their children. They will also send a video of themselves reading with a child, receive text-messages based on these materials as well as the print materials during the last three months of the intervention.
  Interventions: Behavioral: Reading Readiness

INTERVENTIONS:
Behavioral: Healthy Feeding, Healthy Eating — Home Based Motivational Interviewing to Improve Diet Quality of Preschoolers
  Arms: Healthy Feeding, Healthy Eating
Behavioral: Reading Readiness — Active Control that uses Motivational Interviewing to improve Reading Readiness of Preschool Children
  Arms: Reading and Readiness

SUMMARY:
U.S. children eat too little fruits and vegetables and whole grains, and too many energy dense foods, dietary behaviors associated with increased morbidity from cardiovascular diseases. Parents play a key role in shaping their child's diet and best practices suggest that parents should involve children in food preparation, offer, model and encourage a variety of healthy foods. In addition, while parents help to shape food preferences, not all children respond in the same way and certain appetitive traits, such as satiety responsiveness (sensitivity to internal satiety signals), food responsiveness (sensitivity to external food cues), and enjoyment of food may help explain some of these differences. Prior interventions among preschool aged children to improve their diet have not used a holistic approach that fully targets the home food environment, by focusing on food quality, food preparation, and positive feeding practices while acknowledging a child's appetitive traits. This proposal will build upon pre-pilot work to develop and pilot-test the feasibility, acceptability and preliminary efficacy of a novel home-based intervention. The proposed 6-month intervention, will include 3 monthly home visits by a community health worker (CHW) trained in motivational interviewing, that include in-home cooking demos. In between visits, parents will receive tailored text-messages 2x/wk. and monthly mailed tailored materials. During the last 3 months CHW phone calls will replace the home visits. The intervention will be tailored for individual families based on the child's appetitive traits. The proposed research will lay the groundwork for a larger trial to support, motivate, and empower low-income parents to prepare healthy meals and use healthy feeding practices, which will improve children's diets and ultimately their health.

DETAILED DESCRIPTION:
There is a critical need for primary prevention interventions to help parents shape children's dietary behaviors early in life. These interventions need to be convenient for busy, working families and tailored to children's needs and the family environment. Although there have been several interventions among preschool aged children to improve dietary behaviors, none have used a holistic approach that fully targets the home food environment, by focusing on food quality, food preparation, and positive feeding practices while acknowledging a child's appetitive traits. The proposed research will develop and pilot-test the feasibility, acceptability and preliminary efficacy of a novel home-based intervention to improve the diet quality and family food environment of high-risk preschool age, low-income, ethnically diverse children. This research will build upon previous research including a pre-pilot intervention with 15 mother-child dyads which included two home visits: the first visit included a meal-recording and the second included a motivational interviewing (MI) session using coded video clips from the meal-recording as feedback on the parents' feeding practices. All families were retained and significant improvements in several parental feeding practices were found. Based on lessons learned in the pre-pilot, the proposed 6-month intervention will include home visits by a community health worker (CHW) trained in MI, enhanced by adding several innovative components. The home visits will include in-home cooking demonstrations; tailored text-messages, mailed materials and CHW phone calls. The intervention will be tailored for families based on the child's appetitive traits and eating behaviors. These strategies are expected to increase parental knowledge, self-efficacy, and motivation for serving easy, inexpensive healthy foods in the home, leading to increased child exposure to more healthy and varied foods, improvements in parental feeding practices, and ultimately, improvements in child diet quality. The specific aims are as follows:

Aim 1: To conduct focus groups with 40 ethnically diverse low-income parents of preschoolers (2-5 years) to inform the adaptation and development of the enhanced intervention.

Aim 2: To conduct a pilot randomized controlled trial with 60 parent-child pairs (30 intervention/30 control) from ethnically diverse, low-income families with preschoolers to:

Aim 2.1 Determine the feasibility and acceptability of the enhanced intervention.

Aim 2.2 Determine the preliminary efficacy of the enhanced intervention on changes in children's diet quality (primary outcome) and parental feeding practices and availability of healthy foods in the home (secondary outcomes) and calculate effect sizes for a future randomized controlled trial (RCT).

The investigators hypothesize that the intervention will be feasible and acceptable to parents and that parent-child pairs randomized to the intervention condition will demonstrate greater improvements in the outcomes after six months compared to the comparison condition (attention control of a school readiness intervention).

Exploratory aim: Explore how parents' skills, self-efficacy and intrinsic motivation are related to changes in children's diet quality and parental feeding practices.

ELIGIBILITY:
Inclusion Criteria:

* Speak English or Spanish
* Have a child between 2- 5 years of age
* Live with their child most of the time
* Have a phone that is able to video-record
* Be willing to have evening meals video recorded in the home

Exclusion Criteria:

*Has a diagnosed feeding disorder, dietary restrictions, or medical condition that impacts how they feed their child.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fox K, Gans K, McCurdy K, Risica PM, Jennings E, Gorin A, Papandonatos GD, Tovar A. Rationale, design and study protocol of the 'Strong Families Start at Home' feasibility trial to improve the diet quality of low-income, ethnically diverse children by helping parents improve their feeding and food preparation practices. Contemp Clin Trials Commun. 2020 Jun 16;19:100583. doi: 10.1016/j.conctc.2020.100583. eCollection 2020 Sep. PMID 32637721
- [Background] McCurdy K, Gans KM, Risica PM, Fox K, Tovar A. Food insecurity, food parenting practices, and child eating behaviors among low-income Hispanic families of young children. Appetite. 2022 Feb 1;169:105857. doi: 10.1016/j.appet.2021.105857. Epub 2021 Dec 10. PMID 34896386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through a variety of active and passive strategies. For active recruitment, Special Supplemental Nutrition Program for Women, Infants and Children (WIC) nutritionists collected contact information of interested participants, which was then passed to research staff for follow-up. Study staff members also recruited caregivers in WIC waiting rooms or child welfare organizations.
Groups:
- Healthy Feeding, Healthy Eating: The experimental arm will receive three home visits over the first three months of the intervention.Visits will be conducted by a community health worker (CHW) trained in Motivational Interviewing. The home visits will include video-feedback on a meal; in-home cooking demonstrations; tailored text-messages, and mailed materials. During the last three months of the intervention, CHW will conduct monthly phone calls, together with mailed materials and text messages. The intervention will be tailored for families based on the child's appetitive traits and eating behaviors.
  Healthy Feeding, Healthy Eating: Home Based Motivational Interviewing to Improve Diet Quality of Preschoolers
Period: Overall Study
Arm/Group | Healthy Feeding, Healthy Eating | Reading and Readiness
Started | 33 | 30
Completed | 24 | 16
Not Completed | 9 | 14
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Feeding, Healthy Eating | Reading and Readiness | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.67 (6.94) | 34.27 (8.36) | 34.48 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 26 | 55
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 12 | 24
  Multiracial | 6 | 5 | 11
  Unknown | 9 | 6 | 15
  Other | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 33 | 30 | 63
Gender of target child [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 15 | 20 | 35
Caregiver's relationship to child [Count of Participants; unit: Participants]
  Mother | 30 | 27 | 57
  Father or other | 3 | 3 | 6
Country of birth [Count of Participants; unit: Participants]
  United States | 11 | 13 | 24
  Other | 22 | 17 | 39
Language used at home [Count of Participants; unit: Participants]
  English | 9 | 12 | 21
  Spanish | 23 | 18 | 41
  Missing | 1 | 0 | 1
Annual Household Income [Count of Participants; unit: Participants]
  < $25,000 | 14 | 20 | 34
  $25,000-74,999 | 14 | 6 | 20
  >75,000 | 2 | 1 | 3
  Unknown | 3 | 3 | 6
Highest level of education [Count of Participants; unit: Participants]
  Less than 8th grade | 4 | 5 | 9
  High School | 11 | 12 | 23
  College | 18 | 13 | 31
Employment status [Count of Participants; unit: Participants]
  Employment full time | 10 | 5 | 15
  Employment part time | 6 | 7 | 13
  Other, includes employed seasonally, unemployed/looking for work, student, homemaker and disable. ) | 17 | 18 | 35
Marital status [Count of Participants; unit: Participants]
  Married | 15 | 13 | 28
  Not married includes never married, separated, divorced, widowed. | 15 | 10 | 25
  Missing | 3 | 7 | 10
Currently living with a spouse/partner [Count of Participants; unit: Participants]
  Yes | 23 | 20 | 43
  No | 8 | 9 | 17
  Missing | 2 | 1 | 3
Number of other adults living in home [Count of Participants; unit: Participants]
  None | 2 | 3 | 5
  One | 9 | 6 | 15
  Two or more | 21 | 21 | 42
  Missing | 1 | 0 | 1
Number of children (<18 y) living at home [Count of Participants; unit: Participants]
  One | 8 | 11 | 19
  Two or more | 25 | 19 | 44
Currently pregnant [Count of Participants; unit: Participants]
  Yes | 2 | 5 | 7
  No | 27 | 22 | 49
  Missing | 4 | 3 | 7
Food Assistance [Count of Participants; unit: Participants]
  Yes | 27 | 24 | 51
  No | 6 | 5 | 11
  Missing | 0 | 1 | 1
Food insecurity [Count of Participants; unit: Participants]
  Yes, Includes any level of food insecurity | 11 | 17 | 28
  No | 22 | 13 | 35
Target child attends childcare [Count of Participants; unit: Participants]
  Yes | 11 | 9 | 20
  No | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: HEI-2015 Total and Component Scores
Description: HEI-2015 scores will be calculated from twenty four hour recall data (two of them which are combined and scored per 1000 kcal or as a % of intake per NCI scoring guidelines). HEI was designed to measure diet quality in terms of how well diets conform to the 2015 Dietary Guidelines for Americans. The total HEI score represents the sum of 12 components scores (minimum component can be 0 and maximum component score shown in parentheses for each), including total fruit (5), whole fruit (5), total vegetables (5), green and beans (includes dark green vegetables and cooked, dried beans and peas because intakes of these types of vegetables are furthest from the amounts recommended in the USDA Food Patterns) (5), whole grain (10), dairy (10), total protein food (5), seafood and plant proteins (5), fatty acids (10), refined grains (10), sodium (10) added sugar (10), saturated fat (10). Higher scores reflect better outcomes.
Time Frame: Healthy Eating Index Scores at study completion (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Feeding, Healthy Eating | Reading and Readiness
Number analyzed (Participants) | 24 | 16
score on a scale
  HEI-2015 total | 61.6 (10.8) | 65.7 (12.9)
  HEI-2015 Total Vegetable | 2.1 (1.5) | 2.3 (1.5)
  HEI-2015 Greens & Beans | 2.5 (2.4) | 2.7 (2.3)
  HEI-2015 Total Fruit | 3.9 (1.6) | 3.8 (1.8)
  HEI-2015 Whole Fruit | 4.1 (1.7) | 2.8 (2.4)
  HEI-2015 Whole Grain | 4.6 (3.4) | 4.0 (3.9)
  HEI-2015 Total Dairy | 8.3 (2.7) | 8.7 (2.0)
  HEI-2015 Total Protein | 4.5 (1.8) | 4.0 (1.6)
  HEI-2015 Seafood Plant Protein | 2.3 (2.4) | 3.1 (2.2)
  HEI-2015 Fatty Acid | 3.5 (3.1) | 5.2 (3.1)
  HEI-2015 Sodium | 4.8 (3.2) | 7.0 (2.7)
  HEI-2015 Refined Grain | 6.6 (2.9) | 7.0 (2.9)
  HEI-2015 Added Sugar | 7.4 (2.7) | 7.5 (3.2)
  HEI-2015 Saturated Fats | 7.0 (3.1) | 7.6 (3.0)
Statistical Analysis 1: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 total score controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 1.00, Regression, Linear — Familywise error rates were controlled at alpha=.05 for primary and secondary outcomes separately using Holm's sequentially rejective procedure; Slope = -0.55, Standard Error of Mean 4.69
Statistical Analysis 2: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 total vegetable component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 1.00, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -0.35, Standard Error of Mean 0.49
Statistical Analysis 3: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 greens and beans component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 0.20, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = 0.06, Standard Error of Mean 0.88
Statistical Analysis 4: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 total fruit component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 0.20, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = 1.71, Standard Error of Mean 0.67
Statistical Analysis 5: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 whole fruit component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 0.19, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = 2.14, Standard Error of Mean 0.83
Statistical Analysis 6: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 whole grain component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 1.0, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = 0.83, Standard Error of Mean 1.1
Statistical Analysis 7: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 total dairy component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 1.0, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -0.90, Standard Error of Mean 0.85
Statistical Analysis 8: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 total protein foods component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 1.00, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = 0.22, Standard Error of Mean 0.42
Statistical Analysis 9: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 seafood and plant protein component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = -0.12, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -0.12, Standard Error of Mean 0.85
Statistical Analysis 10: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 fatty acid component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 1.00, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -0.31, Standard Error of Mean 1.12
Statistical Analysis 11: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 sodium component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 1.00, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -2.09, Standard Error of Mean 0.97
Statistical Analysis 12: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 refined grains component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 1.00, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -0.80, Standard Error of Mean 1.16
Statistical Analysis 13: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Inverse probability of retention weighted normal linear regression models for between-arm differences in HEI-2015 added sugar component controlling for baseline HEI-2015 saturated fat, child involvement in food preparation, and receipt of any food assistance; Test type: Superiority; p = 1.00, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -0.28, Standard Error of Mean 1.13
Statistical Analysis 14: Comparison: Healthy Feeding, Healthy Eating vs Reading and Readiness; Test type: Superiority; p = 1.00, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -0.52, Standard Error of Mean 0.86

2. Secondary Outcome: Food Parenting Practices
Description: The intervention effects on 14 subscales of the Food Parenting Inventory were used as secondary outcome measures: Encourage try new foods (P), Encourage exploration of new foods (P), Urge child to eat new foods (P), Repeated Presentation of New foods (P), Family meals (P), Regular timing of meals and snacks (P), Inconsistent mealtimes (N), Indifferent feeding (N), Child involvement in food preparation (P), Pressure to Eat (N), Restriction (N), Food as a reward (N), Responsiveness to child's fullness cues (P), Monitoring (P). We also use one subscale of the Comprehensive Feeding Practices Questionnaire: Healthy Eating Guidance (P). All scales are rated on a 5-point Likert scale ranging from 1 (min) to 5 (max). Higher subscale scores indicate greater use of that child feeding practice. We have noted which practice has more positive/desirable practices with a (P) and more negative/not desired sub-scales have an (N) with higher scores.
Time Frame: Food Parenting Practices at study completion (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Feeding, Healthy Eating | Reading and Readiness
Number analyzed (Participants) | 24 | 16
units on a scale
  Encourage try new foods (P) | 4.1 (0.5) | 4.1 (0.6)
  Encourage exploration of new foods (P) | 3.9 (0.9) | 3.9 (1.2)
  Urge child to eat new foods (P) | 4.2 (0.7) | 4.1 (0.8)
  Repeated Presentation of New foods (P) | 4.0 (0.9) | 4.0 (0.9)
  Family meals (P) | 4.4 (0.5) | 3.6 (0.8)
  Regular timing of meals and snacks (P) | 4.3 (0.6) | 2.2 (1.0)
  Inconsistent mealtimes (N) | 2.1 (0.9) | 2.2 (1.0)
  Indifferent feeding (N) | 2.5 (1.2) | 2.7 (1.1)
  Child involvement in food preparation (P) | 3.0 (0.8) | 2.8 (1.2)
  Pressure to Eat (N) | 3.3 (1.1) | 3.4 (1.1)
  Restriction (N) | 4.0 (1.2) | 4.1 (1.1)
  Food as a reward (N) | 3.0 (1.0) | 3.5 (0.9)
  Responsiveness to child's fullness cues (P) | 4.2 (0.8) | 3.6 (1.2)
  Monitoring (P) | 3.8 (1.0) | 3.8 (1.2)
  Healthy Eating Guidance (P | 4.6 (0.4) | 4.4 (0.7)

3. Other Pre Specified Outcome: Home Food Availability Change
Description: Home Food Inventory Change Scores. Home food inventory (HFI) will be used to assess a wide range of commonly available foods in the home environment. A total healthy food availability score will be created from the following items (fruit- frozen, canned, fresh or dried, vegetables-frozen, fresh or canned, milk, water, whole grains, legumes) with a higher score representing more availability of healthy foods. Scores can range from 0-11. An unhealthy food score will also be created from the following items (Chips, Cakes/Cookies, Candy, Pastries, Juice, Soda, Sports drinks, Sweetened Beverages)- scores can range from 0-8 with higher scores representing availability of unhealthy foods.
Time Frame: Changes in Home Food Inventory Scores between baseline and study completion at 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Healthy Feeding, Healthy Eating | Reading and Readiness
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 0/33 | 0/30

LIMITATIONS AND CAVEATS:
In consideration of our study findings, there are some limitations worth noting. First, given the COVID-19 pandemic, several modifications had to be made to the intervention and data collection procedures. We were not able to test our initial fully home-based model and had to modify our secondary outcome of observing changes in the home food environment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Data Collection Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT03923491/Prot_001.pdf
  • Study Protocol: Intervention Delivery Protocol (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03923491/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT03923491/SAP_003.pdf
  • Informed Consent Form (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03923491/ICF_000.pdf